CLINICAL TRIAL: NCT06058936
Title: Effectiveness of Virtual Reality Using Pablo Game Training Program on Upper Extremity Muscle Strength, Pain, Function and Activity of Daily Living in Post-operative Breast Cancer Female Patients.
Brief Title: Exercises Using Virtual Reality on Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoniem Ibrahim, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2023-366
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial with 2 arms parallel design
Who Masked: Outcomes Assessor
Masking Description: Concealed allocation will be performed by a researcher who will not be involved in the treatment of assessment. Permuted blocks will be used to ensure an equal 1:1 allocation ratio. Due to the nature of the study, the assessor and the data analyzer will be blindfolded (double-blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): The patients in this group are under exercise training and pneumatic pressure followed by Pablo©Handle training for 45 minutes per week for 8 week
  -Pablo©Handle training One-dimensional therapy games using five games are available for Pablo©Handle which are (Recycle, Firefighters, Shooting Cans, Balloon, and Apple hunter) The session will be 3 min for each game about 15 min for each session 3 times per week for 8 week
  Interventions: Other: exercises using virtual reality technology
- regular exercises (Active Comparator): The patients in this group will receive exercise training and pneumatic pressure only for 30 min3 times per week for 8 week
  * Exercise training will be done by the following exercise for 15 min3 times per week for 8 week
  * Intermittent Compression Therapy Parameters: using the (Care Pump expert 8)
  * Pressure. 60 mmHg, Direction. Distal to proximal, Speed 4 to 5, for 15 min /3 times per week for 8 week
  Interventions: Other: exercises using virtual reality technology

INTERVENTIONS:
Other: exercises using virtual reality technology — this is a one-dimensional therapy game using (Handle/ or Multiball) five games are available for the Pablo©Handle which are (Recycle, Firefighters, Shooting Cans, Balloon, and Applehunter) The session will be 3 min for each game about 15 min for each session 3 times per week for 8 week
  Other Names: Pablo©Handle training

SUMMARY:
in this study, a randomized controlled trial will be conducted to evaluate the effect of adding exercises using virtual reality on achievements in patients having breast cancer and conducted surgical treatment

DETAILED DESCRIPTION:
in this study, a randomized controlled trial will be conducted to evaluate the effect of adding exercises using virtual reality on achievements in patients having breast cancer and conducted surgical treatment.

A virtual reality (VR) environment is created by combining computer systems and sensor technology with the use of three-dimensional graphics and enabling users to experience a more real, immersive experience by utilizing their various senses (vision, hearing, touch, etc.) through the use of the computer and sensor technologies and it is characterized by immersion, imagination, and interaction 2 groups will be selected randomly to receive experimental and control intervention for 1 month and outcomes will be collected before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer female patients
* Age ≥40 years
* All patients with Eastern Cooperative Oncology Group performance status score ≤ 2
* Having to undergo primary treatment with surgery, chemotherapy, and/or radiotherapy based on the patient's need

Exclusion Criteria:

* Severe anemia (Hb ≤ 8 g/dL)
* Uncontrolled hypertension, diabetes
* severe infection, neurologic or muscular diseases prohibiting physical activity
* severe heart disease or myocardial infarction during the last six months, and a severe chronic obstructive pulmonary disease
* uncontrolled and/or extensive brain metastases, or bone metastases that were assessed to pose a risk of pathological fractures from exercising
* Contraindications given by the physician

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — due to the nature of the study population (breast cancer). only females who suffered breast cancer and underwent surgical treatment will be included
Enrollment: 54 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | at baseline
  will be measured by Pablo system for the affected and unaffected upper limbs
handgrip strength | after the end of the treatment (after 8 weeks)
  will be measured by Pablo system for the affected and unaffected upper limbs
wrist joint active range of motion (ROM) | baseline
  flexion and extension active ROM of the wrist joints will be assessed using Pablo system
wrist joint active ROM | after the end of the treatment (after 8 weeks)
  flexion and extension active ROM of the wrist joints will be assessed using Pablo system
Disabilities of the Arm, Shoulder and Hand (DASH) | at baseline
  DASH is a 30-item questionnaire. Each item is scored on a 1 (no difficulty) to 5 (unable) scale. The total score may range from 0 to 100 points. High scores indicate a high level of disability.
Disabilities of the Arm, Shoulder and Hand (DASH) | after the end of the treatment (after 8 weeks)
  DASH is a 30-item questionnaire. Each item is scored on a 1 (no difficulty) to 5 (unable) scale. The total score may range from 0 to 100 points. High scores indicate a high level of disability.
Fatigue by Multidimensional Fatigue Inventory | at baseline
  The MFI is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue.
Fatigue by Multidimensional Fatigue Inventory | after the end of the treatment (after 8 weeks)
  The MFI is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue.
Anxiety by The State Anxiety Inventory (SAI) | at baseline
  SAI is a valid and commonly used measure for anxiety The SAI includes 20 items; each item is scored on a 4-point Likert scale The SAI range of total scores is between 20 and 80, with the higher score indicating more anxiety
Anxiety by The State Anxiety Inventory (SAI) | after the end of the treatment (after 8 weeks)
  SAI is a valid and commonly used measure for anxiety The SAI includes 20 items; each item is scored on a 4-point Likert scale The SAI range of total scores is between 20 and 80, with the higher score indicating more anxiety
Pain using Numerical Rating Scale (NRS) | at baseline
  this scale is valid and reliable measure of pain intensity. the patient is asked to rate pain intensity be choosing a number from 0 to 10 where 0 indicates no pain and 10 indicates the worst pain ever
Pain using Numerical Rating Scale (NRS) | after the end of the treatment (after 8 weeks)
  this scale is valid and reliable measure of pain intensity. the patient is asked to rate pain intensity be choosing a number from 0 to 10 where 0 indicates no pain and 10 indicates the worst pain ever

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No